CLINICAL TRIAL: NCT07032428
Title: Efficacy of kTMP, a Novel Non-invasive Brain Stimulation Method, for the Treatment of Anhedonia
Acronym: kTMP Anhedonia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Magnetic Tides (Industry)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: Magnetic Tides Inc.
Record Dates: First submitted 2025-06-14; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Anhedonia in Major Depressive Disorder
Keywords: kTMP; NIBS; anhedonia; Major Depressive Disorder; Cortical Excitability; Plasticity; Neuroscience; reward network; kilohertz Transcranial Magnetic Perturbation
MeSH Terms: conditions — Anhedonia; Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active kTMP (Experimental): Participants received 8 V/m of active stimulation
  Interventions: Device: A new non-invasive brain stimulation tool
- Sham kTMP (Sham Comparator): Participants received 0.0 V/m of sham stimulation
  Interventions: Device: A new non-invasive brain stimulation tool with sham setting selected

INTERVENTIONS:
Device: A new non-invasive brain stimulation tool — kTMP is a magnetic induction method that delivers continuous kHz-frequency cortical electric fields (E-fields) which may be amplitude-modulated to potentially mimic electrical activity at endogenous frequencies which will be tested on anhedonia patients in this study.
  Arms: Active kTMP
Device: A new non-invasive brain stimulation tool with sham setting selected — This device will counterbalance the active kTMP conditions
  Arms: Sham kTMP

SUMMARY:
The goal of this proposal is to provide a first assessment of the efficacy of our innovative non-invasive brain stimulation system, kTMP, in the treatment of anhedonia in MDD.

DETAILED DESCRIPTION:
The goal of this clinical trial is to to test and validate a novel, first-in-class, non-invasive approach to engage the brain reward circuitry for treating anhedonia, a core symptom of Major Depressive Disorder (MDD). We've developed a kilohertz Transcranial Magnetic Perturbation (kTMP) device that non-invasively modulates neural activity without patient discomfort. The trial will assess the proof-of-mechanism for kTMP's efficacy in improving anhedonia in MDD patients.

ELIGIBILITY:
Inclusion Criteria: (1) Patients 21-65 years of age with clinically significant anhedonia, as defined by a SHAPS score of at least 20, and (2) Meet DSM-VTR diagnostic criteria for Major Depressive Disorder.

Exclusion Criteria:(1) Reason to anticipate possible hospitalization during the course of the study; (2) Current/history of a psychotic disorder, current manic or mixed episode, meeting the DSM-VTR criteria for bipolar disorder, post-traumatic stress disorder, schizophrenia, at screening, autism spectrum disorders, or mental retardation; (3) Meet DSM-VTR criteria for a substance use disorder within the last year; (4) Current suicidal ideation, suicidal ideation with intent, plan or attempt within the last year, or are considered at significant risk for suicide during the study; (5) Use of any drugs/medications that may interfere/interact with the expected outcomes of the study within 5 half-lives of study participation (see Human Subject section for details); (6) History of seizure; (7) Intracranial expansive process; (8) Pacemaker or any metal implants in head/neck region; (9) Pregnancy; (10) Uncontrolled medical problems including but not limited to severe cardiovascular and cardiopulmonary disease, severe alcohol or drug abuse within the past year; (11) Contraindications for non-invasive brain stimulation or magnetic resonance imaging procedures; (12) Any other condition that in the opinion of the investigator would preclude participation in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2028-07-30 (Estimated); Study Completion 2028-07-30 (Estimated)

PRIMARY OUTCOMES:
Ventral striatal BOLD response during reward anticipation | 2 months
  To assess ventral striatal activation during reward anticipation, patients will participate in a Monetary Incentive Delay (MID) task while in an MRI scanner. We will measure the change in BOLD response during reward anticipation trials, comparing active and sham kTMP and the parametric effect of kTMP on the BOLD response.
The relationship between the level of ventral striatal engagement and clinical scores of anhedonia | 2 months
  For each patient, we will obtain the Snaith-Hamilton Pleasure Scale (SHAPS) scores and carry out a multiple regression analysis

SECONDARY OUTCOMES:
Changes in scores of the Snaith-Hamilton Pleasure Scale (SHAPS). | 6 months
  The Snaith-Hamilton Pleasure Scale (SHAPS) is a well-validated 14-item questionnaire used to assess anhedonia. It asks participants to agree or disagree with statements of hedonic response in pleasurable situations.
The response bias in the Probabilistic Reward Task (PRT). | 6 months
  This task is designed to assess the propensity to modulate behavior as a function of reinforcement history and has been found to reflect reward-related function.
The motivation to pursue reward in the Effort Expenditure for Rewards Task (EEfRT). | 6 months
  The primary outcome measure in EEfRT is the proportion of high-effort, high-reward choices a participant makes with respect to low-effort, low-reward option, which indicates their willingness to expend effort to attain a larger reward.
Scores in the Visual Analog Scale of Anhedonia (VAS). | 6 months
  The Visual Analog Scale (VAS)-Anhedonia is a standard VAS assessment of anhedonia severity which provides a global anhedonia indicator.
Scores in the Temporal Experience of Pleasure Scale (TEPS). | 6 months
  The TEPS is an 18-item self-report measurement of anticipatory and consummatory components of anhedonia which consists of a series of statements that must be rated according to how accurate they are for the individual.
Scores in the Hamilton Rating Scale for Depression (HAM-D). | 6 months
  The HAM-D 17-item version will be included in exploratory analysis to provide confirmatory support for changes in depression severity with treatment.
Scores in the Hamilton Rating Scale for Anxiety (HAM-A). | 6 months
  The HAM-A is a rating scale designed to measure the severity of anxiety symptoms.
Scores in The Cognitive and Physical Functioning Questionnaire | 6 months
  The Cognitive and Physical Functioning Questionnaire (CPFQ) is a 7-item self-report instrument was intended to be a brief scale for measuring cognitive and executive dysfunction in patients with mood and anxiety disorders.
Scores in The Columbia Suicide Severity Rating Scale (CSSRS) | 6 months
  A suicide risk assessment tool that supports suicide risk assessment through a series of simple, plain-language questions that anyone can ask.
Scores in The Clinical Global Impression - Severity (CGI-S) | 6 months
  The CGI-S is a widely administered clinician rated global measure of subject overall illness severity.
Scores in The Clinical Global Impression - Improvement (CGI-I) | 6 months
  The CGI-I is a widely administered clinician rated global measure of the degree of improvement from the initial assessment in subject overall illness severity.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: ELife paper accepted: Kilohertz Transcranial Magnetic Perturbation (kTMP): A New Non-invasive Method to Modulate Cortical Excitability — https://elifesciences.org/reviewed-preprints/92088